CLINICAL TRIAL: NCT04573582
Title: A Phase 1 Open-Label Single-Dose Study to Assess the Pharmacokinetics of Enasidenib (CC 90007) in Subjects With Mild, Moderate and Severe Hepatic Impairment
Brief Title: Pharmacokinetics of Enasidenib (CC-90007) in Participants With Mild, Moderate and Severe Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90007-CP-007; U1111-1257-6808 (Registry Identifier: WHO)
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; CC-90007; Phase 1; Enasidenib
MeSH Terms: interventions — enasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Enasidenib (CC-90007) tablet (Experimental): Participants will receive one 100 mg enasidenib (CC-90007) tablet the morning of Day 1 which will be administered in the fasted state.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — 100 mg enasidenib (CC-90007)
  Other Names: AG-221; AG-221 mesylate; AGI-12910; AGI-12910 mesylate; CC-90007; IDHIFA

SUMMARY:
This is a multi-center, open-label study to assess the PK of single 100 mg oral doses of enasidenib (CC-90007) in subjects with mild, moderate, and severe hepatic impairment (HI), and in matched healthy control subjects with normal hepatic function.

Degrees of hepatic impairment will be determined during screening by the subject's score according to Pugh's Modification of Child's Classification of Severity of Liver Disease.

Subjects will be enrolled in 4 Groups as follows:

* Group A: Approximately 8 subjects with mild hepatic impairment (with a Child-Pugh score of < 7) will be enrolled in Group A.
* Group B: Approximately 8 subjects with moderate hepatic impairment (with a Child-Pugh score of ≥ 7 to ≤ 9) will be enrolled in Group B.
* Group C: Approximately 8 subjects with severe hepatic impairment (with a Child-Pugh score of ≥ 10 to ≤ 15) will be enrolled in Group C.
* Group D: Approximately 8-24 healthy subjects with normal hepatic function will be enrolled in Group D. Subjects in Group D will be matched to subjects in Groups A-C with respect to sex, age (± 10 years), and weight (± 30 pounds). More than 1 subject with differing degrees of HI can be matched to a single control; however, all subjects with HI must be matched to at least 1 healthy match subject.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for all subjects (Groups A, B, C, D) Each subject must satisfy all of the following criteria to be enrolled in the study.

1. Subject must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject is able to communicate with the Investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules and other protocol requirements.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements, including the restrictions.
4. 4. Male, or non-pregnant and non-nursing female between ≥ 40 and ≤ 75 years of age the time of signing the ICF..
5. Body mass index (BMI) ≥ 18 and ≤ 40 kg/m2 at screening.
6. Supine systolic blood pressure (BP): 90 to 160 mmHg, supine diastolic BP:50 to 100 mmHg, and pulse rate: 40 to 100 bpm.
7. Subject is afebrile.
8. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized at least 6 months before screening, or be naturally postmenopausal.
9. Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline Visits. While receiving IP and for at least 2 months after taking the last dose of IP, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options.
10. Male subjects must:

    1. Practice true abstinence or
    2. agree to use a barrier method of birth control during sexual contact with a pregnant female or FCBP while participating in the study, during dose interruptions, and for at least 2 months after the last dose of IP, even if he has undergone a successful vasectomy.

    Inclusion Criteria for Subjects with mild, moderate, or severe hepatic impairment (Groups A-C)

    Each subject with mild, moderate, or severe hepatic impairment must also meet all the applicable criteria listed below for study entry:
11. Subject has moderate or severe hepatic impairment or cirrhosis due to chronic hepatic disease and/or prior alcohol use.
12. Subject has mild (Group A), moderate (Group B), or severe (Group C) hepatic impairment as defined by Child-Pugh Score.

    1. Group A subjects must have mild hepatic impairment and are required to have documentary confirmation of the diagnosis of cirrhosis made by biopsy, laparoscopy, or imaging study with a Child-Pugh score of < 7, at screening.
    2. Group B subjects must have moderate hepatic impairment and are required to have documentary confirmation of the diagnosis of cirrhosis made by biopsy, laparoscopy, or imaging study with a Child-Pugh score of ≥ 7 to ≤ 9, at screening.
    3. Group C subjects must have severe hepatic impairment. If biopsy or laparoscopy is not performed prior to screening, subject can be included only if they have chronic liver disease and objective evidence of portal hypertension (ascites diagnosis by imaging or varices), or current medication for consequences of portal hypertension.

    In either case a Child-Pugh score of ≥ 10 to ≤ 14 at screening is required. Subjects should be enrolled into the group corresponding to the Child-Pugh classification score that most accurately reflects the most severe hepatic disease classification within the past 6 months (based on past medical history or physical examination observation).
13. Must be medically stable for at least 1 month before screening with clinically acceptable medical history, PE, clinical laboratory tests, vital signs, and 12-lead ECGs consistent with the underlying stable mild (Group A), moderate (Group B), or severe (Group C) hepatic impairment condition, as judged by the Investigator.
14. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:

    • Subject (male or female) has a QTcF value ≤ 500 msec at screening.
15. Must be stable on a concomitant medication regimen before dosing with study drug).
16. Subjects may be treated with diuretics for ascites; however, subjects with severe ascites at time of enrollment may only be included at the discretion of the investigator with agreement of the Sponsor.
17. Subjects may have a history of encephalopathy; however, they must be on stable treatment for at least 1 month prior to screening, and must not have had an acute encephalopathic episode in the 1 months prior to screening.

    Inclusion Criteria for a Matched Healthy Subject (Group D)

    Each matched healthy subject must also meet all applicable criteria listed below for study entry:
18. Subject must be free of any clinically significant disease that would interfere with the study evaluations.
19. Subject must have liver-related laboratory test results within the respective reference ranges or with clinically insignificant excursions therefrom as agreed by the Investigator.
20. Subject in Group D must match at least one subject in Groups A-C, as needed with respect to sex, age (± 10 years), and weight (± 30 pounds).
21. Subject must be in good health as determined by past medical history, PE, vital signs, ECG, and clinical laboratory safety tests. Clinical laboratory safety tests (ie, hematology, chemistry, and urinalysis) and 12-lead ECGs must be within normal limits or clinically acceptable as judged by the Investigator.
22. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:
23. If male, subject has a QTcF value ≤ 450 msec at screening;
24. If female, subject has a QTcF value ≤ 470 msec at screening.

Exclusion Criteria:

Exclusion Criteria for all Subjects (Group A, B, C, and D) The presence of any of the following will exclude a subject from enrollment.

1. Subject has any condition or circumstance that prevents the subject from understanding and signing the ICF.
2. Subject has any condition that places the subject at an unacceptable risk from participating in the study or would confound the ability to interpret data from the study.
3. Subject has any significant medical condition or psychiatric illness that would prevent the subject from participating in the study at Investigator discretion.
4. Subject has any surgical or medical condition(s) possibly affecting drug absorption, distribution, metabolism, excretion, eg, bariatric procedure. Subjects with cholecystectomy and appendectomy may be included.

   a. Subject has an estimated creatinine clearance < 60 mL/min as calculated using the Cockcroft-Gault formula- at screening and baseline (Day -1).
5. Subject is pregnant or is breastfeeding.
6. Subject participated in Study CC-90007-CP-003.
7. Subject donated blood or plasma within 2 weeks before dose administration to a blood bank or blood donation center.
8. Subject has a history of alcohol abuse within 6 months before the first dose administration, or positive alcohol screen.
9. Subject has a history of drug abuse within 6 months before the first dose administration, or positive drug screen that is not consistent with the patient's prescribed medication and or/medical history.
10. Subject is known to have active serum hepatitis, or have a positive result to the test for Human immunodeficiency virus (HIV) antibodies at screening.

    • Chronic or resolved Hepatitis B or Hepatitis C are acceptable only if sequelae are limited to hepatic involvement and its consequent comorbidities. (ie, Vasculitis, clinically significant cryoglobulinemia, etc. are unacceptable.)
11. Subject was exposed to an investigational drug within 30 days before dosing, or 5 half-lives of that investigational drug, if known (whichever is longer).
12. Subject used approved medications or herbal medicines that are moderate or strong cytochrome P450 (CYP)1A2, CYP2B6 CYP2C8, CYP2C9, CYP2C19, CYP2D6, and CYP3A4/5 inducers and/or inhibitors (including St. John's wort) within 14 days or 5 half-lives of screening, whichever is longer.
13. Subject will have consumed Seville oranges, grapefruit or grapefruit juice and/or pomelos, exotic citrus fruits, or grapefruit hybrids within 14 days or 5 half-lives of dosing, whichever is longer.
14. Subject smokes more than 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
15. Subject has a history of multiple drug allergies or drug-related anaphylaxis.
16. Subject has received live vaccination (excluding seasonal flu vaccination) within 90 days of dosing.
17. Subject is part of the staff personnel or a family member of the investigational study staff.
18. Subject is, for any reason, deemed by the investigator to be inappropriate for this study, including a subject who is unable to communicate or to cooperate with the investigator or the clinical staff.
19. Subject has had a Transjugular intrahepatic portosystemic shunt (TIPS) procedure.
20. Positive SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) test or signs/symptoms of COVID-19 (Coronavirus Disease 2019) infection.
21. Participants currently in other interventional trials, including those for COVID-19, may not participate in BMS clinical trials until the protocol specific washout period is achieved. If a study participant has received an investigational COVID-19 vaccine or other investigational product designed to treat or prevent COVID-19 prior to screening, enrollment must be delayed until the biologic impact of the vaccine or investigational product is stabilized, as determined by discussion between the Investigator and the Medical Monitor.

    Exclusion Criteria for Subjects with Hepatic Impairment (Group A, B, and C) The presence of any of the following will exclude a hepatically impaired subject from enrollment.
22. Subject has any unstable medical condition occurring within 3 months prior to signing the ICF (excluding hepatic impairment and associated comorbidities per Investigator discretion).
23. Subject has any serious medical condition (excluding hepatic impairment and related complications), clinically significant laboratory abnormality not related to hepatic impairment and related complications, or psychiatric illness that would prevent the subject from signing the ICF and participating in the study per Investigator discretion.
24. Subject has hepatic encephalopathy with time- or place- disorientation, somnolence, stupor, rigidity, coma, no personality/behavior, rigidity, or hyperactive reflexes - or has had such within 1 month of screening.
25. Subject has a history of incipient/planned liver transplantation within 6 months of screening or has received a liver transplant.
26. Subject has a history of hepatorenal syndrome or hemolysis.

    Exclusion Criteria for a Matched Healthy Subject (Group D) The presence of any of the following will exclude a healthy match subject from enrollment.
27. Subject has any clinically significant laboratory abnormality that in the opinion of the Investigator, is considered to prevent the subject from safely completing the study.
28. Subject has any unstable clinically significant illness within 3 months prior to the study.
29. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
30. Positive testing for any active hepatitis, or history of Hepatitis B or C.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-13 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax (CC-90007) | Up to Day 1
  Estimation of maximum observed plasma concentration
Pharmacokinetics - AUC0-∞ (CC-90007) | Up to Day 36
  Estimation of AUC from time zero extrapolated to infinity
Pharmacokinetics - AUC0-t (CC-90007) | Up to Day 36
  Estimation of AUC from time zero extrapolated to last time point
Pharmacokinetics - Tmax (CC-90007) | Up to Day 1
  Time to reach Cmax

SECONDARY OUTCOMES:
Pharmacokinetics - Cmax (AGI-16903) | Up to Day 1
  Estimation of maximum observed plasma concentration
Pharmacokinetics - AUC0-∞ (AGI-16903) | Up to Day 36
  Estimation of AUC from time zero extrapolated to infinity
Pharmacokinetics - AUC0-t (AGI-16903) | Up to Day 36
  Estimation of AUC from time zero extrapolated to last time point
Pharmacokinetics - Tmax (AGI-16903) | Up to Day 1
  Time to reach Cmax
Adverse Events (AEs) | From the time the ICF is signed until Day 36 (+/- 2 days) or within 28 days after the last dose of IP, whichever time frame is longer
  An AE is any noxious, unintended, or untoward medical occurrence that may appear or worsen in a subject during the course of a study. It may be a new intercurrent illness, a worsening concomitant illness, an injury, or any concomitant impairment of the subject's health, including laboratory test values, regardless of etiology. Any worsening (ie, any clinically significant adverse change in the frequency or intensity of a preexisting condition) should be considered an AE.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - Local Institution - 002, Miami, Florida
  - Local Institution - 003, Orlando, Florida
  - Volunteer Research Group and New Orleans Center for Clinical Research - Knoxville, Knoxville, Tennessee

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com